CLINICAL TRIAL: NCT04963803
Title: Improving Aphasia Outcomes Through tDCS-Mediated Attention Management
Brief Title: Improving Aphasia Using Electrical Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R21DC017787-01A1 (NIH); 1R21DC017787-01A1 (NIH)
Record Dates: First submitted 2021-06-21; First posted 2021-07-15 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Aphasia
Keywords: tDCS; attention; language; speech-language therapy
MeSH Terms: conditions — Stroke; Aphasia; Language; Communication Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active transcranial direct current stimulation (tDCS) paired with speech-language therapy (Experimental): Active transcranial direct current stimulation (tDCS) will be delivered using a Soterix mini-CT device. Participants receiving this treatment will be administered 2 milliamperes (mA) of current for 20 minutes/session with the anode electrode placed over F3 and the cathode electrode placed over Fp2 (according to the 1020 system). The tDCS will be paired with 60 minutes of speech-language therapy focusing simultaneously improving auditory comprehension and behavioral attention. All study participants will receive 10 sessions of this combination treatment with no more than one session per day 2-3 times per week.
  Interventions: Device: Active transcranial direct current stimulation (tDCS); Behavioral: Language Specific Attention Treatment
- Sham transcranial direct current stimulation (tDCS) paired with speech-language therapy (Sham Comparator): Sham transcranial direct current stimulation (tDCS) will be delivered using a Soterix mini-CT device. Participants receiving this treatment will be administered 2 milliamperes (mA) of current for 1 minute to simulate the experience of tDCS, after which the current will be ramped down to zero for the remaining 19 minutes of the session with the anode electrode placed over F3 and the cathode electrode placed over Fp2 (according to the 1020 system). The tDCS will be paired with 60 minutes of speech-language therapy focusing simultaneously improving auditory comprehension and behavioral attention. All study participants will receive 10 sessions of this combination treatment with no more than one session per day 2-3 times per week.
  Interventions: Device: Sham transcranial direct current stimulation (tDCS); Behavioral: Language Specific Attention Treatment

INTERVENTIONS:
Device: Active transcranial direct current stimulation (tDCS) — Active transcranial direct current stimulation will be delivered using a Soterix mini-CT device. Participants receiving this treatment will be administered 2 milliamperes (mA) of current for 20 minutes/session for 10 sessions.
  Arms: Active transcranial direct current stimulation (tDCS) paired with speech-language therapy
Device: Sham transcranial direct current stimulation (tDCS) — Sham transcranial direct current stimulation will be delivered using a Soterix mini-CT device. Participants receiving this treatment will be administered 2 milliamperes (mA) of current for 1 minute to simulate the experience of tDCS, after which the current will be ramped down to zero for the remaining 19 minutes of the session. Participants in this arm will receive sham stimulation for 10 sessions.
  Arms: Sham transcranial direct current stimulation (tDCS) paired with speech-language therapy
Behavioral: Language Specific Attention Treatment — This is a specific type of speech-language therapy that focuses on simultaneously improving auditory comprehension and behavioral attention. All study participants will receive 10 sessions of this treatment.

SUMMARY:
Language and communication are essential for almost every aspect of human life, but for people who have aphasia, a language processing disorder that can occur after stroke or brain injury, even simple conversations can become a formidable challenge. Speech and language therapy can help people recover their language ability, but often requires months or even years of therapy before a person is able to overcome these challenges. This research will investigate non-invasive brain stimulation as a way to enhance the effects of speech and language therapy, which may ultimately lead to better and faster recovery from stroke and aphasia. The investigators hypothesize that participants with aphasia who receive speech and language therapy paired with active electrical brain stimulation will improve significantly more on a language comprehension task than those who receive speech and language therapy paired with sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older.
2. No diagnosis of neurological disorder (other than stroke).
3. No diagnosis of psychiatric disorder.
4. No seizure within the past 6 months.
5. Not pregnant.
6. In chronic phase of recovery, defined as at least 6 months post-stroke.
7. Not undergoing speech and language therapy targeting auditory comprehension or attention for the duration of the study.
8. No metal implants in the head.
9. No unhealed skull fractures.
10. Onset of aphasia related to left hemisphere stroke.
11. Damaged brain tissue from stroke does not overlap with left hemisphere dorsolateral prefrontal cortex.
12. Mild to moderate aphasia.
13. Cognitive ability minimally within functional limits.
14. Able to pass vision and hearing screening (with use of corrective aids if needed; eyeglasses, hearing aids).
15. Willing to allow audio-recording of study sessions.

Exclusion Criteria:

1. Younger than 18 years old.
2. Diagnosis or history of neurological disorder other than stroke.
3. Diagnosis or history of psychiatric disorder.
4. History of seizures within the past 6 months.
5. Pregnant.
6. <6 months post-stroke (however, if this is only exclusionary criterion met, participant can be re-evaluated at the 6-month mark if still interested in the study)
7. Currently undergoing speech and language therapy targeting auditory comprehension or attention.
8. Metal implants in the head.
9. Currently has a skull fracture.
10. Onset of aphasia related to etiology other than left hemisphere stroke.
11. Damaged brain tissue includes left hemisphere dorsolateral prefrontal cortex.
12. No aphasia or severe aphasia.
13. Cognitive ability below functional limits.
14. Unable to pass vision and/or hearing screening with use of corrective aids.
15. Unwilling to allow audio-recording of study sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Syracuse University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include self-reported demographic data (e.g., age, race, gender), medical information related to participant's stroke (e.g., date of onset, lesion location), and behavioral data obtained from cognitive and language tasks administered in the Syracuse University Aphasia Lab as part of the study. The final computerized dataset will be stripped of all personal identifiers. The investigators will make the data and associated documentation available to users only via a signed data-sharing agreement that stipulates a commitment to: (1) only use the data for research purposes and not to identify any individual participants, (2) securely storing the data via password-protected databases and secure servers, and (3) destroying or returning the data after analyses are completed. Data sharing will be available upon publication of the main study findings.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 1 year after publication.
Access Criteria: The investigators will make the data and associated documentation available to users only via a signed data-sharing agreement that stipulates a commitment to: (1) only use the data for research purposes and not to identify any individual participants, (2) securely storing the data via password-protected databases and secure servers, and (3) destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Peach RK, Nathan MR, Beck KM. Language-Specific Attention Treatment for Aphasia: Description and Preliminary Findings. Semin Speech Lang. 2017 Feb;38(1):5-16. doi: 10.1055/s-0036-1597260. Epub 2017 Feb 15. PMID 28201833
- [Background] Peach RK, Beck KM, Gorman M, Fisher C. Clinical Outcomes Following Language-Specific Attention Treatment Versus Direct Attention Training for Aphasia: A Comparative Effectiveness Study. J Speech Lang Hear Res. 2019 Aug 15;62(8):2785-2811. doi: 10.1044/2019_JSLHR-L-18-0504. Epub 2019 Jul 25. PMID 31348732
- [Background] Fridriksson J, Rorden C, Elm J, Sen S, George MS, Bonilha L. Transcranial Direct Current Stimulation vs Sham Stimulation to Treat Aphasia After Stroke: A Randomized Clinical Trial. JAMA Neurol. 2018 Dec 1;75(12):1470-1476. doi: 10.1001/jamaneurol.2018.2287. PMID 30128538
- [Background] Riley EA, Wu Y. Artificial grammar learning with transcranial direct current stimulation (tDCS): A pilot study. Brain Stimul. 2019 Sep-Oct;12(5):1307-1308. doi: 10.1016/j.brs.2019.07.002. Epub 2019 Jul 2. No abstract available. PMID 31300247
- [Background] Petersen SE, Posner MI. The attention system of the human brain: 20 years after. Annu Rev Neurosci. 2012;35:73-89. doi: 10.1146/annurev-neuro-062111-150525. Epub 2012 Apr 12. PMID 22524787
- [Background] Woods AJ, Antal A, Bikson M, Boggio PS, Brunoni AR, Celnik P, Cohen LG, Fregni F, Herrmann CS, Kappenman ES, Knotkova H, Liebetanz D, Miniussi C, Miranda PC, Paulus W, Priori A, Reato D, Stagg C, Wenderoth N, Nitsche MA. A technical guide to tDCS, and related non-invasive brain stimulation tools. Clin Neurophysiol. 2016 Feb;127(2):1031-1048. doi: 10.1016/j.clinph.2015.11.012. Epub 2015 Nov 22. PMID 26652115
- [Background] Floel A, Rosser N, Michka O, Knecht S, Breitenstein C. Noninvasive brain stimulation improves language learning. J Cogn Neurosci. 2008 Aug;20(8):1415-22. doi: 10.1162/jocn.2008.20098. PMID 18303984
- [Background] Chhatbar PY, Chen R, Deardorff R, Dellenbach B, Kautz SA, George MS, Feng W. Safety and tolerability of transcranial direct current stimulation to stroke patients - A phase I current escalation study. Brain Stimul. 2017 May-Jun;10(3):553-559. doi: 10.1016/j.brs.2017.02.007. Epub 2017 Feb 27. PMID 28279641
- [Background] Fan J, McCandliss BD, Sommer T, Raz A, Posner MI. Testing the efficiency and independence of attentional networks. J Cogn Neurosci. 2002 Apr 1;14(3):340-7. doi: 10.1162/089892902317361886. PMID 11970796
- [Background] Ishigami Y, Eskes GA, Tyndall AV, Longman RS, Drogos LL, Poulin MJ. The Attention Network Test-Interaction (ANT-I): reliability and validity in healthy older adults. Exp Brain Res. 2016 Mar;234(3):815-27. doi: 10.1007/s00221-015-4493-4. Epub 2015 Dec 8. PMID 26645310
- [Background] Bikson M, Grossman P, Thomas C, Zannou AL, Jiang J, Adnan T, Mourdoukoutas AP, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Jankord R, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Safety of Transcranial Direct Current Stimulation: Evidence Based Update 2016. Brain Stimul. 2016 Sep-Oct;9(5):641-661. doi: 10.1016/j.brs.2016.06.004. Epub 2016 Jun 15. PMID 27372845

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Transcranial Direct Current Stimulation (tDCS) Paired With Speech-language Therapy | Sham Transcranial Direct Current Stimulation (tDCS) Paired With Speech-language Therapy
Started | 12 | 11
Completed | 11 | 11
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Transcranial Direct Current Stimulation (tDCS) Paired With Speech-language Therapy | Sham Transcranial Direct Current Stimulation (tDCS) Paired With Speech-language Therapy | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7) | 63 (12) | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 9 | 5 | 14
Western Aphasia Battery-Revised [Mean (Standard Deviation); unit: Raw score] — Overall score from the Western Aphasia Battery-Revised, also known as the Aphasia Quotient score. Scores from 0-100, higher is less severe.
  Raw score | 80 (20) | 64 (29) | 72 (26)
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 10 | 19
  Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Language Specific Attention Treatment Probe
Description: Measurement of auditory comprehension for untrained sentence-level stimuli. Participants listen to a sentence and are asked to answer comprehension questions about the sentence they heard. Results are reported as the percentage of correct responses out of the total number of items administered. Higher percentages indicate better performance and less auditory comprehension impairment.
Time Frame: Pre-treatment: Baseline measure collected before treatment; Post-treatment: 5-6 weeks after baseline; Follow-up: 10-11 weeks after baseline
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Active Transcranial Direct Current Stimulation (tDCS) Paired With Speech-language Therapy | Sham Transcranial Direct Current Stimulation (tDCS) Paired With Speech-language Therapy
Number analyzed (Participants) | 11 | 11
Percent
  Pre-treatment | 56 (19) | 47 (29)
  Post-treatment | 64 (24) | 52 (29)
  Follow up | 61 (25) | 51 (27)

2. Secondary Outcome: Continuous Performance Test
Description: Change in sustained attention as measured by mean reaction time on the Continuous Performance Test. Participants monitor a screen and press a button for all stimuli except a specific 'no-go' target. The value reported is the mean response time in milliseconds (ms) for correct 'go' trials; a decrease in time indicates improved processing speed.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Active Transcranial Direct Current Stimulation (tDCS) Paired With Speech-language Therapy | Sham Transcranial Direct Current Stimulation (tDCS) Paired With Speech-language Therapy
Number analyzed (Participants) | 11 | 11
ms
  Pre-treatment | 493 (89) | 485 (118)
  Post-treatment | 456 (86) | 507 (133)
  Follow-up | 444 (66) | 529 (158)

3. Secondary Outcome: Attention Network Test
Description: The Attention Network Test (ANT) is a computerized task that measures the efficiency of three distinct attentional networks: Alerting, Orienting, and Executive (Conflict) control.
  Alerting Network Score: Calculated by subtracting the mean reaction time (RT) of double-cue trials from no-cue trials. Range: -500ms to +500ms. Higher positive scores represent a greater alerting benefit.
  Orienting Network Score: Calculated by subtracting the mean RT of spatial-cue trials from center-cue trials. Range: -500ms to +500ms. Higher positive scores represent a greater orienting benefit.
  Conflict (Executive) Network Score: Calculated by subtracting the mean RT of congruent flanker trials from incongruent flanker trials. Range: -500ms to +1000ms. Lower scores represent better executive control and less interference from distracting stimuli.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Active Transcranial Direct Current Stimulation (tDCS) Paired With Speech-language Therapy | Sham Transcranial Direct Current Stimulation (tDCS) Paired With Speech-language Therapy
Number analyzed (Participants) | 11 | 11
ms
  Alerting, pre-treatment | 51 (50) | 43 (76)
  Alerting, post-treatment | 43 (33) | 68 (27)
  Alerting, follow-up | 68 (27) | 60 (30)
  Orienting, pre-treatment | 14 (106) | 14 (36)
  Orienting, post-treatment | 25 (32) | 8 (55)
  Orienting, follow-up | 25 (22) | 29 (32)
  Conflict, pre-treatment | 66 (174) | 123 (96)
  Conflict, post-treatment | 146 (134) | 71 (80)
  Conflict, follow-up | -1 (376) | 76 (61)

4. Secondary Outcome: Scenario Test
Description: The Scenario Test assesses daily life communication and discourse through 6 multi-modal scenarios presented via pictures. Participants are prompted to respond to specific communicative situations. Performance is scored based on the effectiveness of communication (verbal and non-verbal) for each item. Results are reported as the average percentage of correct communicative acts out of the total possible score. Range: 0% to 100%, where higher percentages indicate better functional communication and less severe impairment.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Active Transcranial Direct Current Stimulation (tDCS) Paired With Speech-language Therapy | Sham Transcranial Direct Current Stimulation (tDCS) Paired With Speech-language Therapy
Number analyzed (Participants) | 11 | 11
Percent
  Pre-treatment | 47.5 (6.7) | 44 (13)
  Post-treatment | 48.9 (6.6) | 46 (8)
  Follow-up | 49.2 (6) | 45 (10)

5. Secondary Outcome: Revised Token Test
Description: The Revised Token Test assesses auditory comprehension battery; 5 subtests were administered that contributed to the total score. Results are reported as a mean of the 5 subtest scores. Range of scores is 1 to 15, higher scores represent better performance and less severe auditory comprehension impairment.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scaled score
Arm/Group | Active Transcranial Direct Current Stimulation (tDCS) Paired With Speech-language Therapy | Sham Transcranial Direct Current Stimulation (tDCS) Paired With Speech-language Therapy
Number analyzed (Participants) | 11 | 11
Scaled score
  Pre-treatment | 14 (1) | 13 (2)
  Post-treatment | 14 (1) | 12 (2)
  1-month Follow-up | 14 (1) | 12 (2)

ADVERSE EVENTS:
Time Frame: From enrollment to end of follow-up, 1 month after conclusion of treatment (10-11 weeks)
Arm/Group | Active Transcranial Direct Current Stimulation (tDCS) Paired With Speech-language Therapy | Sham Transcranial Direct Current Stimulation (tDCS) Paired With Speech-language Therapy
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
Study was started in 2021 and COVID significantly affected the ability to recruit and enroll eligible individuals in treatment. Final participant numbers were below our original targets, resulting in underpowered statistical tests.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT04963803/Prot_SAP_ICF_000.pdf